CLINICAL TRIAL: NCT06651905
Title: Superior Laryngeal Nerve Block Versus Sedation with Intravenous Dexmedetomidine Infusion for Awake Fiberoptic Intubation of Hemimandibulectomy Patients with an Anticipated Difficult Airway: a Randomized Controlled Trial
Brief Title: Nerve Block Vs Sedation Infusion for Awake Fiberoptic Intubation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Zayed, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Cairo University, Cairo, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-484-2023
Record Dates: First submitted 2024-10-14; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Superior Laryngeal Nerve Block; Sedation; Dexmedetomidine; Awake Fiberoptic Intubation; Hemimandibulectomy; Anticipated Difficult Airway
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients were given 0.5 mcg/kg of dexmedetomidine over 10 minutes via a syringe pump, followed by a maintenance dose of 0.2-0.7 mcg/kg/hour until the end of intubation based on Hemodynamics.
  Interventions: Drug: Dexmedetomidine
- Superior laryngeal nerve block group (Active Comparator): Patients received an airway nerve block through bilateral superior laryngeal nerve block and trans-tracheal injection for recurrent laryngeal nerve.
  Interventions: Drug: Superior laryngeal nerve block

INTERVENTIONS:
Drug: Dexmedetomidine — The patients were given 0.5 mcg /kg dexmedetomidine over 10 min via syringe pump, followed by 0.2-0.7 mcg/kg/hour until the end of intubation according to hemodynamics.
  Other Names: Sedation arm
  Arms: Dexmedetomidine group
Drug: Superior laryngeal nerve block — The patients received an airway nerve block through bilateral superior laryngeal nerve block and trans-tracheal injection for recurrent laryngeal nerve.
  Other Names: Nerve Block arm
  Arms: Superior laryngeal nerve block group

SUMMARY:
This study compares the efficacy and safety of dexmedetomidine infusion versus superior laryngeal nerve block during awake fiberoptic intubation in hemimandibulectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range ≥ 18 or ≤60.
* Both sexes.
* American Society of Anesthesiologists (ASA) II-III.
* Body mass index:18.5 to 30 kg/m2.
* Hemimandibulectomy patients with an anticipated difficult airway [El-Ganzouri Risk Index (EGRI)>3].

Exclusion Criteria:

* Patient's refusal.
* Known allergy to drugs used in the study.
* Neurological disorders.
* Advanced liver or kidney disease.
* Patient with psychiatric disorders.
* Patient who needs postoperative ICU.
* Airway distortion and cervical spine movement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The intubation score | time from introduction of scope of fibroptic device in the mouth of the patient to the insertion of the endotracheal tube between the vocal cords.Time range of 10 minutes
  The intubation conditions score is assessed based on the following criteria:
  (i) Vocal movement: 1 = open, 2 = moving, 3 = closing, 4 = closed. (ii) Coughing: 1 = none, 2 = slight, 3 = moderate, 4 = severe. (iii) Limb movement: 1 = none, 2 = slight, 3 = moderate, 4 = severe.
  Where The Intubation conditions score is :
  Excellent = 1 when all qualities are excellent. Good = 2 when all qualities are either excellent or good. Poor = 3 when the presence of a single poor quality is noted.

SECONDARY OUTCOMES:
The degree of comfort | time from introduction of scope of fibroptic device in the mouth of the patient to the insertion of the endotracheal tube between the vocal cords. Time range of 10 minutes
  The comfort score was evaluated using a five-point fiberoptic intubation comfort scale: 1 = no reaction, 2 = slight grimace, 3 = heavy grimace, 4 = verbal objection, and 5 = defensive movement of head and hands.
Degree of airway obstruction | time from introduction of scope of fibroptic device in the mouth of the patient to the insertion of the endotracheal tube between the vocal cords Time range of 10 minutes
  The degree of airway obstruction (1 - absent, 2 - requiring neck extension, 3 - requiring jaw thrust) was noted
Heart rate | From one minute before intubation to 10 minutes after intubation
  Heart rate is recorded at 1-minute intervals until intubation is completed, followed by measurements every two minutes until 10 minutes after intubation.
Mean arterial pressure | From one minute before intubation till10 minutes after intubation
  Mean arterial blood pressure is recorded at 1-minute intervals until intubation is completed, followed by measurements every two minutes until 10 minutes after intubation.
Ramsay sedation score | From time of injection of Drugs (Dexetodomidine , Lidocaine) to the patient to 10 minutes after intubation
  Ramsay sedation score was recorded as follows: 1: Awake, agitated or restless or both; 2: Awake, cooperative, oriented, and tranquil; 3: Awake but responds to commands only; 4: Asleep, with a brisk response to a light glabellar tap or loud auditory stimulus.
Patient satisfaction score | From the end of the operation to 24 hours postoperative
  The patient satisfaction score (1-excellent, 2-good, 3-reasonable, 4-poor) was documented.
Incidence of complications | From the end of the operation to 24 hours postoperative
  Adverse events such as bradycardia, hypotension, nausea, vomiting, pruritus, respiratory depression, O2 desaturation, or any other complications were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abd EL Halim Kaddah, MD, Study Director — Professor; Mai M EL Rawas, MD, Principal Investigator — Lecturer
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.